CLINICAL TRIAL: NCT02043327
Title: Simulation-based Training for Colonoscopy: Establishing Criteria for Competency
Brief Title: Simulation Based Training in Colonoscopy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Louise Preisler, MD, Rigshospitalet, Denmark
Other Study IDs: PassFailstudy
Record Dates: First submitted 2014-01-10; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Group Identification
Keywords: Colonoscopy; assessment; certification,; simulation,; standard setting
MeSH Terms: conditions — Social Identification

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Experienced in Colonoscopy: two tests on two different modalities of colonoscopy simulators
- Novices in colonoscopy: Two tests on each of trw colonoscopy simulators

SUMMARY:
The aim of this study is to create simulation-based tests with credible pass/fail-standards for two different fidelities of colonoscopy models

1. virtual reality simulator
2. physical model simulator To create pass/ fail standards for certification

DETAILED DESCRIPTION:
Twenty-five physicians (10 consultants with endoscopic experience and 15 fellows in the first year of fellowship without endoscopic experience) will be tested twice on each of the two different simulator models.

Metrics with discriminatory ability will be identified for both modalities. Reliability will be determined A pass/ fail standard will be determined and the concequences explored.

ELIGIBILITY:
Inclusion Criteria: For the two groups

Experienced endoscopists :

Having performed >350 colonoscopy procedures

Novice endoscopists:

First or second year of fellowship in gastroenterology Having performed less than 3 colonoscopies

Exclusion Criteria: For the two groups

Experienced endoscopists:

Prior simulator training

Novice endoscopists:

Prior simulator training

Ages: 28 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Experienced: 10 consultants of gastroenterology with experience in Colonoscopy (>350 procedures) Novices: 15 fellows of gastroenterology with limited experience in Colonoscopy (<2 procedures)
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Metrics with discriminatory ability measuring colonoscopy competence | tests were carried out in one day per participant
  Each participant perform two tests on each model within the same day.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Preisler, MD, Principal Investigator — Rigshospitalet, Copenhagen, University of Copenhagen
Locations (1):
- Rigshospitalet; CEKU, Copenhagen, Copenhagen, Denmark